CLINICAL TRIAL: NCT06454825
Title: Effects of Combined Antiemetic Protocol For The Prevention Of Postoperative Nausea And Vomiting In Orthognathic Surgery: A Randomized Double Blinded Clinical Study
Brief Title: Effects of Antiemetic Agents in Orthognathic Surgery Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Özge Özyılmaz, Associate Professor, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ozgedoganay.001
Record Dates: First submitted 2024-06-01; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Emesis, Postoperative; Maxillofacial Abnormalities
Keywords: anti-emetic agent; orthognathic surgery; granisetron; metoclopramide
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Maxillofacial Abnormalities | interventions — Infusion Pumps

STUDY DESIGN:
Intervention Model Description: randomized double blinded clinical study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Granisetron group (Active Comparator): one group received granisetron 3 mg drug
  Interventions: Drug: Intravenous drug
- Granisetron and Metoclopramide group (Experimental): one group received a combination of granisetron 3 mg and metoclopramide 10 mg drugs
  Interventions: Drug: Intravenous drug

INTERVENTIONS:
Drug: Intravenous drug — medications were applied intravenously to the groups 30 minutes before end of the procedure

SUMMARY:
In an effort to prevent or treat consistently high rates of PONV following maxillofacial operations, several medications, techniques and multimodal protocols have been studied. In the present study, the investigators hypothesized that combining metoclopramide with granisetron will improve PONV incidence when compared with granisetrone alone.

DETAILED DESCRIPTION:
Despite advances in anesthetic techniques and antiemetic drugs that accompany increasing awareness of anesthesia providers, postoperative nausea and vomiting (PONV) remains one of the most common problems after general anesthesia. PONV is one of the major problems leading to patient dissatisfaction, prolonged stay in postoperative care unit and hospital, readmissions and thus it can increase health care costs. In the studies performed in PONV prone patients and high-risk surgeries, as compared with other antiemetic medications, "setrons" provided lower nausea and vomiting incidence postoperatively, but were unable to completely prevent this "big little" problem.The blood in the stomach has been indicated as one of the major causes of PONV following maxillofacial surgery thus, using metoclopramide may relieve the complaints by evacuating this irritant. After institutional ethic committee and National Medicines, 66 consecutive patients, classified as ASA I and II physical status and aged between 18 and 60 years were included in the study. Apfel's simplified PONV risk score including female sex, history of motion sickness or PONV, smoking status and predicted use of postoperative opioids was recorded.Procedures were performed under general anesthesia. Patients in Group G received 3 mg granisetron (Neoset, Deva, Istanbul) and the patients in group GM received 3 mg granisetron + 10 mg metoclopramide (Metpamid, Sifar İlaç, Istanbul) 30 minutes before the end of operation intravenously. A nursing staff collected the data concerning PONV, VAS, systolic, diastolic and mean arterial pressures, heart rate, peripheral arterial saturation, total doses of drugs used, overall bleeding score, infused fluid volume, VAS, surgical procedure, duration of surgery and rescue antiemetics for nausea if applied for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing orthognathic surgery
* ASA I and II physical status
* aged between 18 and 60 years
* must be volunteer to take study drugs

Exclusion Criteria:

* Unable or unwilling to give informed consent
* Underwent to genioplasty
* Documented hypersensitivity to study drugs
* Gastroesophageal reflux or hiatal hernia
* Diabetes mellitus
* Renal insufficiency
* Pregnancy
* Electrolyte imbalance
* Neurological disease
* Mental retardation
* Prolonged QT interval.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting | fully awake and on the 1st, 2nd, 4th, 6th , 8th and 24th hours postoperatively
  The primary outcome of interest in the present study was the incidence of PONV.

SECONDARY OUTCOMES:
Visual analogue scale | fully awake and on the 1st, 2nd, 4th, 6th , 8th and 24th hours postoperatively
  Visual analogue scale was used to record pain score. following the surgery. 0-10 point scale was used. 0 showed no pain, 10 showed worst pain status.
Systolic arterial pressure | preoperatively, at the induction, every 30 minutes interval till the end of the surgery, before extubation.
  It was measured during the surgery.
Diastolic arterial pressure | preoperatively, at the induction, every 30 minutes interval till the end of the surgery, before extubation.
  It was measured during the surgery.
Mean arterial pressure | preoperatively, at the induction, every 30 minutes interval till the end of the surgery, before extubation.
  It was measured during the surgery.
heart rate | preoperatively, at the induction, every 30 minutes interval till the end of the surgery, before extubation.
  It was measured during the surgery.
peripheral arterial saturation | preoperatively, at the induction, every 30 minutes interval till the end of the surgery, before extubation.
  It was measured during the surgery.
total doses of drugs | before extubation
  It was recorded during the surgery.
Bleeding amount | before extubation
  It was recorded at the end of the surgery.
Infused fluid volume | before extubation
  It was recorded during the surgery.
Duration of surgery | before extubation
  It was recorded at the end of the surgery.
Rescue antiemetic | it was recorded until follow-up period ended and if applied it would be recorded. Between fully awake in ward and 24th hours postoperatively.
  It was recorded at the end of the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: ÖZGE 3 ÖZYILMAZ, DDS, Principal Investigator — Bezmialem Vakif University, Faculty of Dentistry
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Patients were anonymously recorded. Due to the data and patient's security, if it requested from the investigators, in that case we will decide.